CLINICAL TRIAL: NCT04436796
Title: The International Diabetes Closed Loop (iDCL) Trial: A Randomized Crossover Comparison of Adaptive Model Predictive Control (MPC) Artificial Pancreas Versus Sensor Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS) in the Outpatient Setting in Type 1 Diabetes (DCLP4)
Brief Title: The International Diabetes Closed Loop (iDCL) Trial: Protocol 4
Acronym: DCLP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G200047; UC4DK108483 (NIH)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas; Automated Insulin Delivery; Closed Loop Control; Continuous Glucose Monitor (CGM); interoperable Artificial Pancreas System (iAPS)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Artificial Pancreas (Experimental): Subjects will be provided the Interoperable Artificial Pancreas System (iAPS) which includes the iAPS phone platform, a study insulin pump, study continuous glucose monitor (CGM), and a study glucometer. This iAPS is designed to help control blood sugar in people living with type 1 diabetes.
  Interventions: Device: interoperable Artificial Pancreas System (iAPS)
- Sensor Augmented Pump/Predictive Low Glucose Suspend (Active Comparator): Subjects will continue use of home insulin pump with a study continuous glucose monitor (CGM) and study glucometer. Subject may use home pump in PLGS mode if this is supported and compatible with the study sensor.
  Interventions: Other: Sensor-Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS)

INTERVENTIONS:
Device: interoperable Artificial Pancreas System (iAPS) — Use of the iAPS at home for 13 weeks, with weekly adaptation of insulin delivery settings occurring automatically in the iAPS.
  Arms: Artificial Pancreas
Other: Sensor-Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS) — Use of personal pump with study CGM & glucometer at home for 13 weeks.
  Arms: Sensor Augmented Pump/Predictive Low Glucose Suspend

SUMMARY:
The investigators aim to compare the efficacy and safety of an AID system using an adaptive MPC algorithm versus SAP (which may or may not include PLGS; to be referred to as SAP) in people with type 1 diabetes.

DETAILED DESCRIPTION:
A randomized crossover trial will compare the efficacy and safety of an automated insulin delivery (AID) study system using an adaptive Model Predictive Control (MPC) algorithm versus SAP (which may or may not include PLGS; to be referred to as SAP) therapy in people with type 1 diabetes for 13 weeks in each arm of the study. A Pilot Phase using the study system for 10-14 days will be conducted prior to the crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
* Using an insulin pump for at least 3 months (which may include use of automated features)
* Familiarity and use of a carbohydrate ratio for meal boluses
* Age ≥18.0 years old
* For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
* If using a personal CGM, willingness to use a Dexcom G6 CGM and discontinue personal CGM use during the study
* Willing not to begin use of, or not to continue use of if currently using, a personal AID (closed loop control) system during the study; note if the system offers an open-loop mode or can be switched to a PLGS mode that is compatible with the Dexcom G6, the system may be used during the study in these modes only
* Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
* Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial, and not to use Afrezza during the trial
* Investigator believes that the participant can successfully and safely operate all study devices and is capable of adhering to the protocol

Exclusion Criteria:

* Use of Afrezza or any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas) unless participant is willing to discontinue during the trial.
* Two or more episodes of DKA requiring an emergency room visit or hospitalization in the past 6 months
* Two or more episodes of severe hypoglycemia with seizure or loss of consciousness in the last 6 months
* Hemophilia or any other bleeding disorder
* A medical or other condition that in the opinion of the investigator could create a safety concern for the participant or put the study at risk. History of frequent severe hypoglycemia or history of frequent severe hyperglycemia and/or ketosis, without emergency room visit or hospitalization, due to poor diabetes self-management may be disqualifying per investigator judgment
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Dassau, PhD, Study Chair — Harvard University; Jordan Pinsker, MD, Study Chair — Sansum Diabetes Research Institute; Francis J Doyle III, PhD, Principal Investigator — Harvard University
Locations (5):
- United States (5):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Stanford University, Stanford, California
  - Joslin Diabetes Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
NIH's Data Sharing Policy on sharing research resources for research purposes to the scientific community will be followed. Data will be stored in a Data Archive Database includes CGM-insulin delivery time series & boluses, will be deidentified & retrievable only by subject ID number. Individual patterns of demographic & insulin treatment parameters leave open a remote possibility of deductive disclosure of subjects with unusual characteristics. Thus, data will be made available only under a Data-Sharing Agreement that includes: (1) a commitment to using the data only for research purposes & not to identify participants; (2) a commitment to securing the data using appropriate computer technology; & (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The dataset from each iDCL protocol will be made public after publication of all manuscripts written by the study group using the dataset and any regulatory submission/completion of review by the regulatory agency, but no later than 3 years after the completion of the protocol even if additional manuscripts or regulatory submissions are planned.

REFERENCES:
- [Result] Pinsker JE, Dassau E, Deshpande S, Raghinaru D, Buckingham BA, Kudva YC, Laffel LM, Levy CJ, Church MM, Desrochers H, Ekhlaspour L, Kaur RJ, Levister C, Shi D, Lum JW, Kollman C, Doyle FJ; iDCL Trial Research Group. Outpatient Randomized Crossover Comparison of Zone Model Predictive Control Automated Insulin Delivery with Weekly Data Driven Adaptation Versus Sensor-Augmented Pump: Results from the International Diabetes Closed-Loop Trial 4. Diabetes Technol Ther. 2022 Sep;24(9):635-642. doi: 10.1089/dia.2022.0084. Epub 2022 Jun 2. PMID 35549708

RESULTS

PARTICIPANT FLOW:
Groups:
- Artificial Pancreas First, Then Sensor-Augmented Pump/Predicitive Low Glucose Suspend: Subjects will be provided the Interoperable Artificial Pancreas System (iAPS) which includes the iAPS phone platform, a study insulin pump, study continuous glucose monitor (CGM), and a study glucometer. This iAPS is designed to help control blood sugar in people living with type 1 diabetes.
  interoperable Artificial Pancreas System (iAPS): Use of the iAPS at home for 13 weeks, with weekly adaptation of insulin delivery settings occurring automatically in the iAPS.
  Subjects will then continue use of home insulin pump with a study continuous glucose monitor (CGM) and study glucometer. Subject may use home pump in PLGS mode if this is supported and compatible with the study sensor.
  Sensor-Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS): Use of personal pump with study CGM & glucometer at home for 13 weeks.
- Sensor Augmented Pump/Predictive Low Glucose Suspend First, Then Artificial Pancreas: Subjects will then continue use of home insulin pump with a study continuous glucose monitor (CGM) and study glucometer. Subject may use home pump in PLGS mode if this is supported and compatible with the study sensor.
  Sensor-Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS): Use of personal pump with study CGM & glucometer at home for 13 weeks.
  Then subjects will be provided the Interoperable Artificial Pancreas System (iAPS) which includes the iAPS phone platform, a study insulin pump, study continuous glucose monitor (CGM), and a study glucometer. This iAPS is designed to help control blood sugar in people living with type 1 diabetes.
  interoperable Artificial Pancreas System (iAPS): Use of the iAPS at home for 13 weeks, with weekly adaptation of insulin delivery settings occurring automatically in the iAPS.
Period: Overall Study
Arm/Group | Artificial Pancreas First, Then Sensor-Augmented Pump/Predicitive Low Glucose Suspend | Sensor Augmented Pump/Predictive Low Glucose Suspend First, Then Artificial Pancreas
Started | 19 | 16
Completed | 19 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Artificial Pancreas First, Then Sensor-Augmented Pump/Predictive Low Glucose Suspend: Subjects will be provided the Interoperable Artificial Pancreas System (iAPS) which includes the iAPS phone platform, a study insulin pump, study continuous glucose monitor (CGM), and a study glucometer. This iAPS is designed to help control blood sugar in people living with type 1 diabetes.
  interoperable Artificial Pancreas System (iAPS): Use of the iAPS at home for 13 weeks, with weekly adaptation of insulin delivery settings occurring automatically in the iAPS.
  After 13 weeks, participants then crossed over to the other arm.
- Sensor Augmented Pump/Predictive Low Glucose Suspend First, Then Artificial Pancreas: Subjects will continue use of home insulin pump with a study continuous glucose monitor (CGM) and study glucometer. Subject may use home pump in PLGS mode if this is supported and compatible with the study sensor.
  Sensor-Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS): Use of personal pump with study CGM & glucometer at home for 13 weeks.
  After 13 weeks, participants then crossed over to the other arm.
- Total: Total of all reporting groups
Arm/Group | Artificial Pancreas First, Then Sensor-Augmented Pump/Predictive Low Glucose Suspend | Sensor Augmented Pump/Predictive Low Glucose Suspend First, Then Artificial Pancreas | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (16) | 37 (15) | 39 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 19 | 10 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percent CGM Time in Range 70-180 mg/dL
Description: This results shown is mean percent time in range 70-180 mg/dL.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 69 (14) | 66 (14)

2. Primary Outcome: Non-inferiority for CGM Time <54 mg/dL
Description: Superiority for time in range 70-180 mg/dL and non-inferiority for time <54 mg/dL measured with CGM will be considered primary endpoints, analyzed using a hierarchical gatekeeping testing procedure
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 0.41 (0.39) | 0.71 (0.82)

3. Secondary Outcome: CGM Mean Glucose
Description: CGM-measured mean glucose (mg/dL)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
mg/dL | 158 (22) | 156 (27)

4. Secondary Outcome: CGM Time > 180
Description: CGM time > 180 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 29 (15) | 30 (16)

5. Secondary Outcome: CGM Time > 250
Description: CGM time > 250 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 9 (8) | 8 (8)

6. Secondary Outcome: CGM Time < 70
Description: CGM time < 70 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 2.1 (1.7) | 3.5 (3.1)

7. Secondary Outcome: CGM Time < 54 (Superiority)
Description: CGM time < 54 mg/dL (Superiority)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 0.41 (0.39) | 0.71 (0.82)

8. Secondary Outcome: Coefficient of Variation
Description: CGM measured glucose variability measured with the coefficient of variation (CV)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage SD of Mean
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage SD of Mean | 34.5 (5.3) | 34.9 (5.7)

9. Secondary Outcome: CGM Time in Range 70-140 mg/dL
Description: CGM-measured % in range 70-140 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 44 (14) | 43 (17)

10. Secondary Outcome: Standard Deviation
Description: CGM measured glucose variability measured with the standard deviation (SD)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
mg/dL | 34.5 (5.3) | 34.9 (5.7)

11. Secondary Outcome: CGM Time < 60
Description: CGM time < 60 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 0.81 (0.73) | 1.39 (1.45)

12. Secondary Outcome: LBGI
Description: Low blood glucose index (LBGI) by CGM with higher index indicating higher risk of hypoglycemia. LBGI ≤ 1.1 is associated with minimal risk of hypoglycemia, 1.1 < LBGI ≤ 2.5 is associated with a low risk of hypoglycemia, 2.5 < LBGI ≤ 5.0 is associated with a moderate risk of hypoglycemia, and LBGI > 5.0 is associated with high risk of hypoglycemia.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
index score | 0.6 (0.4) | 1.0 (0.8)

13. Secondary Outcome: CGM Time > 300
Description: CGM time > 300 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of time | 3 (4) | 3 (4)

14. Secondary Outcome: HBGI
Description: High Blood Glucose Index (HBGI) is a measure of Hyperglycemic Risk based on frequency and severity of hyperglycemic events. HBGI < 4.5 is associated with lower risk of hyperglycemia, 4.5 < HBGI < 9 is associated with a moderate risk of hyperglycemia and HBGI > 9 is associated with high risk of hyperglycemia
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
index score | 6.8 (3.6) | 6.8 (4.1)

15. Secondary Outcome: HbA1c at 13 Weeks
Description: Hemiglobin A1c measured after completing each study arm
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
percentage of glycated hemoglobin | 6.8 (0.8) | 6.8 (0.9)

16. Secondary Outcome: Number of Participants With HbA1c <7.0% at 13 Weeks
Description: Number of participants HbA1c <7.0% after completing each study arm
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
Participants | 19 | 22

17. Secondary Outcome: Number of Participants With HbA1c <7.5% at 13 Weeks
Description: Number of participants HbA1c <7.5% after completing each study arm
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
Participants | 26 | 28

18. Secondary Outcome: Diabetes Distress Scale at 13 Weeks - Total Score
Description: Diabetes Distress Scale for adults has 28 items rated on a 6 point Likert scale that ranges from 1 (not a problem) to 6 (a very serious problem). The total score is the mean of the sum of responses and ranges from 1 to 6 where a higher score indicates greater degrees of diabetes distress.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 34 | 35
score on a scale | 1.6 (0.5) | 1.6 (0.5)

19. Secondary Outcome: Glucose Monitoring Satisfaction Survey (Total Scale)
Description: The GMSS for Type 1 Diabetes contains four subscales as well as a total scale. For this measure, total scale is reported. To calculate the total scale (higher scores indicate greater satisfaction): Mean of all items 1-15 (reverse code items: 2-7, 9, 11-13, and 15) which are all scored on a 5 point scale (1-5) (Minimum Total Scale Score is 1, Maximum Total Scale Score is 5)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 34 | 35
score on a scale | 3.9 (0.8) | 4.0 (0.6)

20. Secondary Outcome: Hypoglycemia Confidence Scale
Description: Hypoglycemia Confidence Scale has 20 items which are rated on a 4-point Likert Scale ranging from 1 (not confident at all) to 4 (very confident) with higher scores indicating higher confidence in dealing with hypoglycemia. A single score is computed by calculating the mean of the sum of all items and ranges from 1 to 4.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 34 | 35
score on a scale | 3.4 (0.5) | 3.5 (0.5)

21. Secondary Outcome: INSPIRE Survey Scores - Following Study System Period Only
Description: The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems: Perceptions, Ideas, Reflections, Expectations (INSPIRE). Survey total scores are computed by calculating the mean of the sum of all item ratings then multiplying the mean by 25 to scale the score to a range from 0 to 100. Higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The Adult survey has 22 items, the Teens/Adolescents survey has 17 items and the Parent survey has 21 items.
Time Frame: 13 weeks
Population: following study system period only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 34 | 0
score on a scale | 67.7 (23.9) |

22. Secondary Outcome: SUS Survey Scores - Following Study System Period
Description: System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicate better perceived usability
Time Frame: 13 weeks
Population: following study system period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 34 | 0
score on a scale | 60.7 (25.5) |

23. Secondary Outcome: Total Daily Insulin
Description: Total Daily Insulin (units)
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: units/kg
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
units/kg | 0.52 [0.43 to 0.68] | 0.52 [0.42 to 0.68]

24. Secondary Outcome: Basal: Bolus Insulin Ratio
Description: Basal: bolus insulin ratio
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
Number analyzed (Participants) | 35 | 35
ratio | 0.99 [0.64 to 1.94] | 1.13 [0.84 to 1.85]

25. Other Pre Specified Outcome: CGM Metrics by Time of Day
Description: Calculate all CGM metrics listed above (including the primary outcome) for: All 24 hours of the day, Daytime only (06:00AM to 00:00AM), Nighttime only (00:00AM to 06:00AM).
Time Frame: 13 weeks
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Number of Participants With Severe Hypoglycemia (Per Protocol)
Description: Severe hypoglycemia (per protocol)
Time Frame: 13 weeks
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Number of Participants With Diabetic Ketoacidosis (Per Protocol)
Description: Diabetic ketoacidosis (per protocol)
Time Frame: 13 weeks
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Ketone Events Defined as Day With Ketone Level >1.0 mmol/L
Description: Ketone events defined as day with ketone level >1.0 mmol/L
Time Frame: 13 weeks
Reporting Status: Not Posted

29. Other Pre Specified Outcome: CGM-measured Hypoglycemic Events (>15 Minutes With Glucose Concentration <54 mg/dL)
Description: CGM-measured hypoglycemic events (>15 minutes with glucose concentration <54 mg/dL) in each arm.
Time Frame: 3 months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: CGM-measured Hyperglycemic Events (>15 Minutes With Glucose Concentration >300 mg/dL)
Description: CGM-measured hyperglycemic events (>15 minutes with glucose concentration >300 mg/dL) in each arm.
Time Frame: 3 months
Reporting Status: Not Posted

31. Other Pre Specified Outcome: BG-measured Hypoglycemic Events (One BG Record <54 mg/dL
Description: BG-measured Hypoglycemic Events (One BG Record <54 mg/dL
Time Frame: 13 weeks
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Worsening of HbA1c From Baseline to 26 Weeks by >0.5%
Description: Worsening of HbA1c from baseline to 26 weeks by >0.5%
Time Frame: 13 weeks
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Other Serious Adverse Events (SAE) and Serious Adverse Device Events (SADE)
Description: Other serious adverse events (SAE) and serious adverse device events (SADE)
Time Frame: 13 weeks
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Adverse Device Effects (ADE)
Description: Adverse device effects (ADE)
Time Frame: 13 weeks
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Unanticipated Adverse Device Effects (UADE)
Description: Unanticipated adverse device effects (UADE)
Time Frame: 13 weeks
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Number of Participants With SH Events
Description: For this outcome, mean +/- SD or summary statistics appropriate to the distribution will be tabulated by treatment group
Time Frame: 13 weeks
Reporting Status: Not Posted

37. Other Pre Specified Outcome: SH Event Rate Per 100 Person-years
Description: For this outcome, severe hypoglycemia event rate per 100 person-years will be calculated as a rate.
Time Frame: 13 weeks
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Number of Participants With DKA Events
Description: For this outcome, number of participants with diabetic ketoacidosis (DKA) will be tabulated.
Time Frame: 13 weeks
Reporting Status: Not Posted

39. Other Pre Specified Outcome: DKA Event Rate Per 100 Person-years
Description: For this outcome, the diabetic ketoacidosis event rate per 100 person-years will be calculated as a rate.
Time Frame: 13 weeks
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Any Adverse Event Rate Per 100 Person-years
Description: For this outcome, the adverse event rate per 100 person-years calculated as a rate.
Time Frame: 13 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From protocol entry through last study date which is approximately 26-28 weeks per participant.
Description: Definitions are the same as the clinicaltrials.gov definition. Please see clinical protocol for exclusions to adverse event collection.
Arm/Group | Artificial Pancreas | Sensor Augmented Pump/Predictive Low Glucose Suspend
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35
Other Adverse Events (participants affected / at risk) | 4/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Pancreas (N=35) | Sensor Augmented Pump/Predictive Low Glucose Suspend (N=35)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Pancreas (N=35) | Sensor Augmented Pump/Predictive Low Glucose Suspend (N=35)
Hyperglycemia or ketosis events without meeting criteria for Diabetic Ketoacidosis (Endocrine disorders) | 4 (4) | 0 (0)
Medical Device Site Bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04436796/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04436796/SAP_001.pdf
  • Informed Consent Form (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT04436796/ICF_002.pdf